CLINICAL TRIAL: NCT01447264
Title: Comparison of the Effectiveness Between Land and Water Exercises on Isokinetic Muscle Strength of Lower Limbs in Women With Rheumatoid Arthritis: a Randomized Controlled Trial
Brief Title: Effectiveness of Water Exercises on Isokinetic Muscle Strength
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Department of Medicine (Ambiguous)
Responsible Party: Principal Investigator, Marcelo M Pinheiro, Clinical Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUSaoPaulo-01
Record Dates: First submitted 2011-10-03; First posted 2011-10-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Muscle strength; Body composition; Physical activity; Water exercises; Hydrotherapy; Randomized controlled clinical trial
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Land exercises (Placebo Comparator): The patients of this group will perform the same exercises from water exercises
  Interventions: Procedure: Land exercises
- Water exercises (Active Comparator): The patients of this group will perform the same exercises from land exercises
  Interventions: Procedure: Water exercises
- Control group (No Intervention): No intervention will be recommended

INTERVENTIONS:
Procedure: Land exercises — 3 times a week. 50 minutes in every session. Performed by educational professor
  Arms: Land exercises
Procedure: Water exercises — 3 times a week. 50 minutes in every session. Performed by educational professor
  Arms: Water exercises

SUMMARY:
The interest in studying the impact of aquatic exercise on muscle strength of patients with rheumatoid arthritis came after publication of several studies that pointed to the potential benefit of exercise on the natural history of the disease, including reduction of pain, better immune response as well as aerobic fitness and functional capacity and increase muscle strength, endurance and quality of life.

In general, the aquatic exercises are indicated for patients with chronic joint diseases, since the aquatic environment seems to be more secure for this population due to the reduction of joint loading, as well as gain range of motion.

However, there are some difficulties to show the real and consistent beneficial effect of physical activity in these patients, such as the small number of randomized controlled clinical trials, short intervention period (4-8 weeks), lack of details of the exercise protocols used, methodological problems (heterogeneous measures to evaluate the outcome, change of medication). Moreover, no study evaluated the disease activity, according to the tool most used clinically worldwide, the DAS28.

It is known that aquatic exercises without impact in healthy subjects are sufficient to gain muscle strength. Nonetheless, in people with joint limitation the benefits from these same exercises to gain muscle strength is not known.

To date, no studies addressing the effect of aquatic exercise on muscle strength and disease activity in patients with rheumatoid arthritis. In addition, there is the need to obtain a standardized protocol for prescribing of aquatic exercises. The choice of lower-limb strength was based on its relevance to the acceleration and deceleration during the march, as well as to perform activities of daily living, leisure and professional in these individuals.

Thus, this study aims at:

1. Exercises performed in the aquatic environment and without the concomitant use of overhead equipment are sufficient to promote gain muscle strength in the lower limb?
2. What is the isolated effect of water resistance on muscle strength? Could it work as an impact that is used in exercises done on the land?

DETAILED DESCRIPTION:
The investigators objectives are:

* To compare the peak torque of flexor and extensor of the knee between land and water exercises in women with rheumatoid arthritis. This is a randomized controlled clinical trial with 16 weeks of length;
* To verify the changes of disease activity, functional capacity and body composition measurements before and after the intervention

ELIGIBILITY:
Inclusion Criteria:

* Females;
* Pre- or postmenopausal;
* Disease Activity: from mild to moderate, according to the DAS28;
* Functional class I and II Steinbrocker;
* No rehabilitation program in the last three months;
* Stable medication in the three months before randomization;
* Cardiorespiratory fitness after exercise testing and cardiologic exam;
* Agree and sign the Instrument of Consent;

Exclusion Criteria:

* Circulatory problems, ulcers in the legs, or other untreated skin lesions that would preclude the exercise in the pool;
* Physical activity regularly in the three months prior to intervention;
* Use of orthoses or any other devices;
* Hip or knee prosthesis;
* Regular use of proteic supplements or anabolic drugs;
* Orthopedic surgery scheduled for the next six months;
* Intra-articular infiltration in the three months prior to randomization or scheduled for the next six months;
* Illiteracy and cognitive impairment;
* Hearing loss and visual;
* Phobia of water;
* Hypersensitivity to the chlorine;
* Epilepsy and urinary or fecal incontinence;
* Any uncontrolled chronic illness.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 16 weeks
  Isokinetic muscle strength

SECONDARY OUTCOMES:
Disease Activity Score (DAS28) | 16 weeks
  To evaluate the disease activity in rheumatoid arthritis
Health Assessment Questionnaire (HAQ) | 16 weeks
  To measure the impact of funcional capacity in patients with rheumatoid arthritis
Body composition measurements | 16 weeks
  Measures of body composition (lean and fat mass), by Dual-X ray absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo M Pinheiro, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil